CLINICAL TRIAL: NCT00004015
Title: Postoperative Treatment of Glioblastoma With BNCT at the Petten Irradiation Facility
Brief Title: Boron Neutron Capture Therapy Following Surgery in Treating Patients With Glioblastoma Multiforme Removed During Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-11961; EORTC-11961
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — mercaptoundecahydrododecaborate; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: sodium borocaptate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Boron neutron capture therapy may selectively kill tumor cells without harming normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of boron neutron capture therapy following surgery in treating patients with glioblastoma multiforme removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine systemic and local toxicity of borocaptate sodium with boron neutron capture therapy (BNCT) following craniotomy with gross total resection in patients with glioblastoma multiforme.
* Determine the qualitative and quantitative dose-limiting toxicity and maximum tolerated dose of this regimen in these patients.
* Determine the maximum tolerated radiation dose of BNCT in cranial localization to healthy tissues in these patients under defined conditions.

OUTLINE: This is a dose escalation, multicenter study.

Within 6 weeks of surgery, patients receive borocaptate sodium followed 12-18 hours later by neutron irradiation. Treatment repeats daily for 4 days.

Cohorts of 3-9 patients receive escalating doses of neutron irradiation. The maximum tolerated dose is defined as the dose preceding that at which 3 or more patients experience dose limiting toxicity.

Patients are followed weekly for 4 weeks, monthly for 2 months, every 6 weeks for 15 months and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 30-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven glioblastoma multiforme for which conventional radiotherapy would be of little or no benefit
* Gross total resection of tumor confirmed by postoperative MRI performed within 48 hours of surgery
* Evaluable preoperative and postoperative MRI films with and without contrast must be available
* No prior brain malignancy
* No prior craniotomy except for glioblastoma

PATIENT CHARACTERISTICS:

Age:

* 50 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin, SGOT, SGPT, and alkaline phosphatase no greater than 2.5 times normal unless caused by reversible reaction to antiseizure medication

Renal:

* Blood urea nitrogen and creatinine no greater than 2.5 times upper limit of normal

Cardiovascular:

* No severe heart disease (e.g., congestive heart failure, angina pectoris)

Pulmonary:

* No severe dyspnea at time of diagnosis
* No severe obstructive or restrictive lung disease

Other:

* No other concurrent malignant tumor
* No severe gastrointestinal disease or active peptic ulcer disease
* No uncontrolled endocrine disease
* No serious mental disease, organic brain disease (e.g., preexisting epilepsy or serious aphasia), or legally incapacitated patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for glioblastoma multiforme
* No concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy for glioblastoma multiforme
* No concurrent chemotherapy

Endocrine therapy:

* No prior endocrine therapy for glioblastoma multiforme except corticosteroids
* No concurrent endocrine therapy

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy for glioblastoma multiforme
* No prior radiotherapy to head and neck
* No other concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior stereotactic biopsy allowed for glioblastoma multiforme

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2002-06; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Acute toxicity as measured by NCIC-Common Toxicity Criteria up to 30 days after the first BSH administration

SECONDARY OUTCOMES:
Late toxicity as measured by RTOC and EORTC late radiation morbidity scale from 90 days after completion of irradiation treatment until death
Overall survival as measured by Logrank until death

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Sauerwein, MD, PhD, Study Chair — Universitaetsklinikum Essen
Locations (8):
- Karl-Franzens-University Graz, Graz, Austria
- Toronto Sunnybrook Regional Cancer Centre at Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Hopital Pasteur, Nice, France
- Germany (2):
  - Universitaetsklinikum Essen, Essen
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
- Ospedale Santa Chiara Pisa, Pisa, Italy
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - EC Joint Research Centre - Institute for Energy, Petten

REFERENCES:
- [Background] Wittig A, Moss RL, Stecher-Rasmussen F, Appelman K, Rassow J, Roca A, Sauerwein W. Neutron activation of patients following boron neutron capture therapy of brain tumors at the high flux reactor (HFR) Petten (EORTC Trials 11961 and 11011). Strahlenther Onkol. 2005 Dec;181(12):774-82. doi: 10.1007/s00066-005-1433-4. PMID 16362787
- [Background] Verbakel WF, Hideghety K, Morrissey J, Sauerwein W, Stecher-Rasmussen F. Towards in vivo monitoring of neutron distributions for quality control of BNCT. Phys Med Biol. 2002 Apr 7;47(7):1059-72. doi: 10.1088/0031-9155/47/7/305. PMID 11996055
- [Background] Husing J, Sauerwein W, Hideghety K, Jockel KH. A scheme for a dose-escalation study when the event is lagged. Stat Med. 2001 Nov 30;20(22):3323-34. doi: 10.1002/sim.954. PMID 11746321
- [Background] Rassow J, Stecher-Rasmussen F, Voorbraak W, Moss R, Vroegindeweij C, Hideghety K, Sauerwein W. Comparison of quality assurance for performance and safety characteristics of the facility for Boron Neutron Capture therapy in Petten/NL with medical electron accelerators. Radiother Oncol. 2001 Apr;59(1):99-108. doi: 10.1016/s0167-8140(00)00298-x. PMID 11295213
- [Background] Sauerwein W, Moss R, Rassow J, Stecher-Rasmussen F, Hideghety K, Wolbers JG, Sack H. Organisation and management of the first clinical trial of BNCT in Europe (EORTC protocol 11961).EORTC BNCT study group. Strahlenther Onkol. 1999 Jun;175 Suppl 2:108-11. doi: 10.1007/BF03038906. PMID 10394415
- [Background] Gabel D, Philipp KH, Wheeler FJ, Huiskamp R. The compound factor of the 10B(n,alpha)7Li reaction from borocaptate sodium and the relative biological effectiveness of recoil protons for induction of brain damage in boron neutron capture therapy. Radiat Res. 1998 Apr;149(4):378-86. PMID 9525503
- [Background] Pignol JP, Oudart H, Chauvel P, Sauerwein W, Gabel D, Prevot G. Selective delivery of 10B to soft tissue sarcoma using 10B-L-borophenylalanine for boron neutron capture therapy. Br J Radiol. 1998 Mar;71(843):320-3. doi: 10.1259/bjr.71.843.9616243.
- [Result] Verbakel WF, Sauerwein W, Hideghety K, Stecher-Rasmussen F. Boron concentrations in brain during boron neutron capture therapy: in vivo measurements from the phase I trial EORTC 11961 using a gamma-ray telescope. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):743-56. doi: 10.1016/s0360-3016(02)04392-4. PMID 12573762
- [Result] Hideghety K, Sauerwein W, Haselsberger K, Grochulla F, Fankhauser H, Moss R, Huiskamp R, Gabel D, de Vries M. Postoperative treatment of glioblastoma with BNCT at the petten irradiation facility (EORTC protocol 11,961). Strahlenther Onkol. 1999 Jun;175 Suppl 2:111-4. doi: 10.1007/BF03038907. PMID 10394416
- [Result] Gabel D, Touw D, Stecher-Rasmussen F, et al.: Quality control of Na2B12H11SH, a drug boron neutron capture therapy in EORTC trial 11961. [Abstract] Ann Oncol 9(suppl 2): 129, 1998.
- [Result] Hideghety K, Sauerwein W, Wittig A, Gotz C, Paquis P, Grochulla F, Haselsberger K, Wolbers J, Moss R, Huiskamp R, Fankhauser H, de Vries M, Gabel D. Tissue uptake of BSH in patients with glioblastoma in the EORTC 11961 phase I BNCT trial. J Neurooncol. 2003 Mar-Apr;62(1-2):145-56. doi: 10.1007/BF02699941. PMID 12749710
- [Result] Hideghety W, Sauerwein W, DeVries M, et al.: Post-operative treatment of glioblastoma with boron neutron capture therapy at the European High Flux Reactor Petten (EORTC protocol 11961). [Abstract] Ann Oncol 9(suppl 2): 129, 1998.
- [Result] Sauerwein W, Hideghety K, De Vries M, et al.: Boron neutron capture therapy (BNCT) for the treatment of glioblastoma (EORTC protocol 11961). [Abstract] Radiother Oncol 48(suppl 1): s157, 1998.
- [Result] Sauerwein W, Hideghety K, De Vries M, et al.: Conducting phase I clinical trial in binary treatment modality: methodical questions for the evaluation of boron neutron capture therapy. [Abstract] Ann Oncol 9(suppl 2): 129, 1998.
- [Result] Vos MJ, Turowski B, Zanella FE, Paquis P, Siefert A, Hideghety K, Haselsberger K, Grochulla F, Postma TJ, Wittig A, Heimans JJ, Slotman BJ, Vandertop WP, Sauerwein W. Radiologic findings in patients treated with boron neutron capture therapy for glioblastoma multiforme within EORTC trial 11961. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):392-9. doi: 10.1016/j.ijrobp.2004.06.008. PMID 15667958
- [Result] Haselsberger K, Pendl G, Sauerwein W, et al.: BNCT for glioblastoma in Europe: design of the EORTC protocol 11961 and clinical course of the first patient. [Abstract] J Neurooncol 39 (2): A-P155, 147, 1998.